CLINICAL TRIAL: NCT06366984
Title: Comparison of Outcome of Plastibell Circumcision Method With Open Surgical Technique in Infants Presenting at Tertiary Care Hospital
Brief Title: Outcome of Plastibell Circumcision Versus Open Method Circumcision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children Hospital and Institute of Child Health, Lahore (Other)
Responsible Party: Principal Investigator, Muhammad Adeel Ashiq, Principal Investigator, Children Hospital and Institute of Child Health, Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Adeel4
Record Dates: First submitted 2024-04-08; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Bleeding; Site Infection
Keywords: Circumcision,; Infection; Bleeding,; Plastibell,
MeSH Terms: conditions — Hemorrhage; Infections

STUDY DESIGN:
Intervention Model Description: Randomized controll trial
Who Masked: Outcomes Assessor
Masking Description: outcome assessor is unaware of group allocated
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plastibell group (Experimental): plastibell method applied for circumcision
  Interventions: Other: plastibell
- open method circumcision (Experimental): open method of circumcision applied
  Interventions: Other: open method

INTERVENTIONS:
Other: plastibell — plastibell used for circumcision
  Arms: Plastibell group
Other: open method — open method used for circumcision
  Arms: open method circumcision

SUMMARY:
To compare the outcomes of plastibell circumcision method with open surgical technique in infants presenting at tertiary care hospital.

Methods This randomized controlled trial (NCT??) was conducted at Pediatric surgery department, the Children's hospital and the University of Child health, Lahore. Study was carried out over a period of six months from 11-01-2022 to 11-07-2022. Non probability, purposive sampling was used. 174 infants presenting for circumcision were admitted and assigned a method of circumcision randomly. They were randomly divided in to 2 groups by using opaque sealed envelope technique. Infants in group A were underwent plastibell circumcision while infants in group B were underwent open technique circumcision. 87 circumcisions were performed by each method. The informed consent was taken from parents for inclusion into the study. All infants were underwent circumcision under local anesthesia as per assigned method. Same preoperative, per-operative, and postoperative care was given to each regardless of the technique. These patients were followed for 3 hours to assess bleeding as per operational definition. Then followed on an outpatient basis every 6th day until complete healing is achieved (30 days).The data regarding age, weight, duration of procedure, wound infection and post circumcision bleeding was recorded in a predesigned performa. (As per operational definition).

DETAILED DESCRIPTION:
Circumcision is a surgical method in which surgical removal of the prepuce (foreskin) is done. Religious, cultural, medical, and common public health reasons are known to be the major indications for this procedure. It is usually done in neonatal age but can also be performed at any age. The WHO has begun to recommend circumcision on the basis of studies indicating its positive effects on human health and especially its role in protection from AIDS. As with adult circumcision, neonatal circumcision may be helpful to reduce the risk of acquiring HIV infection, phimosis and paraphimosis in future adult life. Though Circumcision is one of the commonest procedures in the surgery, still a gold standard approach is not defined. In Pakistan most circumcisions are done in neonatal or infant life, or circumcised in the adult age group. It is a relatively simple procedure with healing time up to 2 weeks.

There are many advantages of male circumcision at younger age than older, which include lower risk of complications, lower cost, and faster healing. Different techniques are being in practice like Plastibell method, Mogen Clamp, bone cutter technique and Free-hand open surgical method.

This randomized control trial was conducted at Pediatric Surgery Department, The Children's Hospital and University of Child Health Sciences, Lahore from 11-01-2022 to 11-07-2022. After approval from the ethical review committee of the hospital, all infants came for circumcision were included except those who need redo circumcision or have Inadequate clinical record or have hypospadias or who are syndromic children.

174 infants presenting for circumcision were admitted and assigned a method of circumcision randomly. They were randomly divided in to 2 groups by using opaque sealed envelope technique. Infants in group A were underwent plastibell circumcision while infants in group B were underwent open technique circumcision. 87 circumcisions were performed by each method. The informed consent was taken from parents for inclusion into the study. All infants were underwent circumcision under local anesthesia as per assigned method. Same preoperative, per-operative, and postoperative care was given to each regardless of the technique. These patients were followed for 3 hours to assess bleeding as per operational definition. Then followed on an outpatient basis every 6th day until complete healing is achieved (30 days).The data regarding age, weight, duration of procedure, wound infection and post circumcision bleeding was recorded in a predesigned performa. (As per operational definition).

The data was entered in SPSS version 23 and analyzed through it. Means and SD was calculated for quantitative variables like age, weight and operation time. Frequency and percentage was calculated for qualitative variables like bleeding and wound infection. Outcomes i.e bleeding and wound infection were compared between both groups by using Chi-square test. P-value ≤ 0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* all uncircumcised male

Exclusion Criteria:

* hypospadias, syndromic children

Ages: 1 Day to 12 Months | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 174 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
infection | 30 days
  incidence of surgical site infection according to southampton score

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad A Ashiq, M.S, Principal Investigator — The Children hospital
Locations (1):
- The Children Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
no plan of sharing